CLINICAL TRIAL: NCT03746587
Title: Multicentre Double-blinded, Randomized Placebo-controlled Study of Arimoclomol in Patients Diagnosed With Gaucher Disease Type 1 or 3
Brief Title: Study of Arimoclomol in Patients Diagnosed With Gaucher Disease Type 1 or 3
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-19 pandemic made it impossible to assess the trial objective
Sponsor: ZevraDenmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OR-ARI-GAU-01
Record Dates: First submitted 2018-11-01; First posted 2018-11-19 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Gaucher Disease, Type 1; Gaucher Disease, Type 3
Keywords: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — arimoclomol

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded, randomized, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arimoclomol I (Experimental): Arimoclomol, oral capsule
  Interventions: Drug: Arimoclomol
- Arimoclomol II (Experimental): Arimoclomol, oral capsule
  Interventions: Drug: Arimoclomol
- Arimoclomol III (Experimental): Arimoclomol, oral capsule
  Interventions: Drug: Arimoclomol
- Placebo (Placebo Comparator): Placebo oral capsule matching experimental arm
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Arimoclomol — Arimoclomol in 3 different dosages
  Arms: Arimoclomol I; Arimoclomol II; Arimoclomol III
Drug: Placebo oral capsule — Matching placebo capsule
  Arms: Placebo

SUMMARY:
Multicenter, doubleblinded, randomized placebo-controlled study of arimoclomol in patients with Gaucher Disease Type 1 or 3

DETAILED DESCRIPTION:
Evaluating the response of 3 dose levels of arimoclomol on various pharmacodynamic biomarkers in blood and cerebrospinal fluid as indicators of enhanced GBA in Gaucher Disease Type 1 or 3.

ELIGIBILITY:
Key Inclusion Criteria:

* Be able to understand and voluntarily sign informed consent
* A diagnosis GD, either Type 1 or Type 3
* For GD3 at least 1 neurological symptom
* Age ≥ 4 years and ≤ 60 years at the time of enrolment
* Plasma or serum chitotriosidase activity greater than 3 times the upper limit of normal.

Key Exclusion Criteria:

* Recipient of a liver transplant or planned liver transplantation during the course of the study.
* Splenectomy within 4 months of study entry or planned splenectomy during the course of the study.
* Severe liver damage.
* Severe renal insufficiency.
* Body weight < 10 kg.

Other inclusion and exclusion criteria may apply

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | 6 months
  The percentage change in serum chitotriosidase levels from baseline to 6 months

SECONDARY OUTCOMES:
Growth Endpoint | 6 months
  Change in weight curve (Khadilkar and Khadilkar, 2011) measured in kilograms, at every 6 months
Growth Endpoint | 6 months
  Change in length curve (Khadilkar and Khadilkar, 2011) measured in meters at every 6 months
Maturation Endpoint | 6 months
  Age at pubertal onset (Tanner Stage II) for subjects who had not reached puberty at screening
Maturation Endpoint | 6 - 12 months
  Tanner Staging at baseline, 6 months and at least every 12 months (Tanner stage I-IV)
Imaging Endpoint | 6 months
  Change in size of liver and spleen assessed by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Aabha Nagral, MD, Principal Investigator — Jaslok Hospital and Reseach Centre, Mumbai
Locations (8):
- India (8):
  - King Edward Memorial Hospital, Mumbai, Maharashtra
  - Jaslok Hospital and Reseach Centre, Mumbai, Maharashtra
  - KEM HOSPITAL Research Centre, Pune, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Christian Medical College and Hospital., Vellore, Tamil Nadu
  - Institute of Child Health, Kolkata, West Bengal
  - Maulana Azad Medical College, New Delhi
  - All India Institute of Medical Sciences, New Delhi

IPD SHARING:
Plan to Share IPD: Undecided